CLINICAL TRIAL: NCT03182543
Title: Physiological Response to Ataulfo Mango Pulp and Peel Beverages in Exercise
Brief Title: Physiological Effect of Ataulfo Mango (Manguifera Indica) Beverage in Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Ciudad Juarez (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UACJ-ICB-2017-01
Record Dates: First submitted 2017-05-29; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Exercise-induced Oxidative Stress
Keywords: Exercise; Oxidative stress; Antioxidant
MeSH Terms: conditions — Motor Activity | interventions — Water

STUDY DESIGN:
Intervention Model Description: The prescription of the treatments (AM1, AM2) and control (water) was randomized. The subject consumed 600mL of AM1, AM2 or water. 2 hours later subject performed the exercise test. Next treatment was evaluated after a week of wash-out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AM1 (Experimental): Mango pulp beverage
  Interventions: Dietary Supplement: Mango pulp beverage
- AM2 (Experimental): Mango pulp and peel beverage
  Interventions: Dietary Supplement: Mango pulp and peel beverage
- Control (Placebo Comparator): Control beverage
  Interventions: Dietary Supplement: Control beverage

INTERVENTIONS:
Dietary Supplement: Mango pulp beverage — The subject consumes mango pulp beverage (200 g mango pulp + 600 mL water). 2 hours later subject performs the exercise test.
  Washout: 1 week washout period prior to the administration of this intervention to avoid possible carryover effect.
  Other Names: AM1; 200 g mango pulp + 600 mL water
  Arms: AM1
Dietary Supplement: Mango pulp and peel beverage — The subject consumes mango pulp and peel beverage (160 g mango pulp + 40 g mango peel + 600 mL water). 2 hours later subject performs the exercise test.
  Washout: 1 week washout period prior to the administration of this intervention to avoid possible carryover effect.
  Other Names: AM2; 160 g mango pulp + 40 g mango peel + 600 mL water
  Arms: AM2
Dietary Supplement: Control beverage — The subject consumes control beverage (600 mL water). 2 hours later subject performs the exercise test.
  Washout: 1 week washout period prior to the administration of this intervention to avoid possible carryover effect.
  Other Names: 600 mL water
  Arms: Control

SUMMARY:
The aim of this study is to assess the antioxidant capacity of two mango base beverages (AM1, AM2), against exercise-induced oxidative stress.

DETAILED DESCRIPTION:
Introduction. The post-consumption physiological effect of mango cv. "Ataulfo" pulp (MP) and peel (MC) in humans before exercise has been poorly evaluated.

Objective. To evaluate the physiological response, to consumption of two mango base beverages, AM1 (200g MP/ 600mL water) and AM2 (160g MP; 40g MC / 600mL water), before and after a submaximal exercise test.

Methods. The antioxidant profile and physicochemical characteristics of AM1 and AM2 were evaluated. Several cardiorespiratory, anthropometric and body composition parameters of 19 university students, prior to the consumption of AM1, AM2 and water, were evaluated in three non-consecutive sessions (self-control cases). The glycemic, lactic and antioxidant (FRAP), uric acid (AU), reduced glutathione (GSH) and lipid oxidation (TBARS) and protein carbonyls (PC) responses were evaluated in plasma before and after an incremental cycle ergometer exercise test.

ELIGIBILITY:
Inclusion Criteria:

* healthy male
* university student
* no alcohol, cigar or drugs consumption

Exclusion Criteria:

* no antioxidant supplement or ergogenic consumption
* health issues with performing physical activity

Ages: 17 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Antioxidant capacity change | 0 min (before beverage intake), 9-15 min (immediately after exercise test)
  Assessed by FRAP change. Blood samples were drawn from the antecubital vein into EDTA test tubes at rest, before beverage intake, and immediately following the exercise test. Samples were then centrifuged at 5000 rpm for 10 min at 4°C to obtain plasma, which was withdrawn and separated into eppendorf vials, maintained at -80°C until further biochemical analysis.
Antioxidant capacity change | 0 min (before beverage intake), 9-15 (immediately after exercise test)
  Assessed by uric acid concentration change. Blood samples were drawn from the antecubital vein into EDTA test tubes at rest, before beverage intake, and immediately following the exercise test. Samples were then centrifuged at 5000 rpm for 10 min at 4°C to obtain plasma, which was withdrawn and separated into eppendorf vials, maintained at -80°C until further biochemical analysis.
Antioxidant capacity change | 0 min (before beverage intake), 9-15 (immediately after exercise test)
  Assessed by reduced glutathione concentration change. Blood samples were drawn from the antecubital vein into EDTA test tubes at rest, before beverage intake, and immediately following the exercise test. Samples were then centrifuged at 5000 rpm for 10 min at 4°C to obtain plasma, which was withdrawn and separated into eppendorf vials, maintained at -80°C until further biochemical analysis.

SECONDARY OUTCOMES:
Oxidative stress change | 0 min (before beverage intake), 9-15 (immediately after exercise test)
  Assessed by TBARS concentration change. Blood samples were drawn from the antecubital vein into EDTA test tubes at rest, before beverage intake, and immediately following the exercise test. Samples were then centrifuged at 5000 rpm for 10 min at 4°C to obtain plasma, which was withdrawn and separated into eppendorf vials, maintained at -80°C until further biochemical analysis.
Oxidative stress change | 0 min (before beverage intake), 9-15 (immediately after exercise test)
  Assessed by protein carbonyls concentration change. Blood samples were drawn from the antecubital vein into EDTA test tubes at rest, before beverage intake, and immediately following the exercise test. Samples were then centrifuged at 5000 rpm for 10 min at 4°C to obtain plasma, which was withdrawn and separated into eppendorf vials, maintained at -80°C until further biochemical analysis.
Lactic acid concentration change | 0 min (before performing exercise test), 3 min, 6 min, 9 min, 12 min, 15 min (during exercise test)
  Assessed by lactic acid concentration change. Capillary blood samples were taken from the fingertip, using a lancet and analyzed (YSI modelo 1500, Yellow Springs, USA)
Postprandial glycemic change | 0 min (before beverage intake), 30 min, 60 min, 90 min, 120 min (after beverage intake)
  Assessed by blood glucose concentration change. Capillary blood samples were taken from the fingertip, using a lancet, and analyzed (ReliOn Confirm/micro Test Strips ARKRAY, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Wall-Medrano, PhD, Study Director — Universidad Autónoma de Ciudad Juárez; Gregorio Chavez-Treviño, MS, Principal Investigator — Universidad Autónoma de Ciudad Juárez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez-Parrilla E, De La Rosa LA, Legarreta P, Saenz L, Rodrigo-Garcia J, Gonzalez-Aguilar GA. Daily consumption of apple, pear and orange juice differently affects plasma lipids and antioxidant capacity of smoking and non-smoking adults. Int J Food Sci Nutr. 2010 Jun;61(4):369-80. doi: 10.3109/09637480903514041. PMID 20109132
- [Background] Ramos-Jimenez A, Hernandez-Torres RP, Wall-Medrano A, Torres-Duran PV, Juarez-Oropeza MA, Solis Ceballos JA. Acute physiological response to indoor cycling with and without hydration; case and self-control study. Nutr Hosp. 2013 Sep-Oct;28(5):1487-93. doi: 10.3305/nh.2013.28.5.6698. PMID 24160205
- [Background] Spirlandeli AL, Deminice R, Jordao AA. Plasma malondialdehyde as biomarker of lipid peroxidation: effects of acute exercise. Int J Sports Med. 2014 Jan;35(1):14-8. doi: 10.1055/s-0033-1345132. Epub 2013 Jun 14. PMID 23771832
- [Background] Wang CY, Haskell WL, Farrell SW, Lamonte MJ, Blair SN, Curtin LR, Hughes JP, Burt VL. Cardiorespiratory fitness levels among US adults 20-49 years of age: findings from the 1999-2004 National Health and Nutrition Examination Survey. Am J Epidemiol. 2010 Feb 15;171(4):426-35. doi: 10.1093/aje/kwp412. Epub 2010 Jan 15. PMID 20080809
- [Background] Wall-Medrano A, Olivas-Aguirre FJ, Velderrain-Rodriguez GR, Gonzalez-Aguilar A, de la Rosa LA, Lopez-Diaz JA, Alvarez-Parrilla E. [Mango: agroindustrial aspects, nutritional/functional value and health effects]. Nutr Hosp. 2014 Nov 1;31(1):67-75. doi: 10.3305/nh.2015.31.1.7701. Spanish. PMID 25561099